CLINICAL TRIAL: NCT01029899
Title: Phase II Study of Evaluation of Handheld Colonoscopy Force Monitor by Expert and Trainee Endoscopists in the Performance of Colonoscopy
Brief Title: Characterize Differences in Force Patterns Used by Different Endoscopists and Trainee Endoscopists
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Georgetown University (Other); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: CFM-05; 2R44DK068936 (NIH)
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Compare Performance of Colonoscopists
Keywords: Colonoscopy; Force; Monitor; Endoscopist; Trainee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is to evaluate how doctors in training are different from very experienced doctors when using force to perform colonoscopy with a device that monitors the amount of force applied to the colonoscope during colonoscopy.

DETAILED DESCRIPTION:
The study consists of two sequential observational studies designed to identify which instrument should be used to assess trainee performance and to quantify trainee skill development in performance of colonoscopy over the course of their training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic or screening colonoscopy ASA Class I or II
* All ethnic and racial groups will be included
* Able to comprehend, sign and date the written informed consent form (ICF)
* English is their primary language

Exclusion Criteria:

* Chronic pathology that in the opinion of the endoscopist could interfere with the colonoscopy. Examples include: colonic stricture, poor preparation, obstructing tumor
* Specific pathology that would limit the extent of examination
* ASA class 3 or greater
* Pregnancy
* Vulnerable subjects. Students, nursing home residents, institutionalized patients, and those with psychological or physical incapacity

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult male and female patients between the ages of 30 and 75 presenting for screening or diagnostic colonoscopy to be performed by any of the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2009-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Colonoscopy Force Monitoring demonstrates patterns of how doctors in training are different from very experienced doctors when they do colonoscopy. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Armen Sarvazyan, Ph.D., D.Sc., Study Chair — Artann Laboratories
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - The University of Washington, Seattle, Washington

REFERENCES:
- [Result] Korman LY, Brandt LJ, Metz DC, Haddad NG, Benjamin SB, Lazerow SK, Miller HL, Greenwald DA, Desale S, Patel M, Sarvazyan A. Segmental increases in force application during colonoscope insertion: quantitative analysis using force monitoring technology. Gastrointest Endosc. 2012 Oct;76(4):867-72. doi: 10.1016/j.gie.2012.05.030. Epub 2012 Jul 27. PMID 22840291